CLINICAL TRIAL: NCT07182838
Title: Conducting an Initial Small, Controlled Clinical Pharmacology Trial to Assess for Therapeutic Biologics Activity (Proof-of-Concept) That Suggests the Potential for Clinical Benefits of HIV (+) Patients
Brief Title: Proof-of-Concept Clinical Pharmacology Trial for HIV Antigen Presentation Therapeutic Biologic Mix
Acronym: HIVGP-BCG
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Collaborators: UnitedHealthcare (Other)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IORG Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IND 179135 Research; FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); IRB00009424 (Registry Identifier: HHS, IRB); IORG0007849 (Registry Identifier: HHS, IORG); NPI-1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI-1023387701 (Registry Identifier: HHS, Health Care Provider Organization); IND 179135 (Registry Identifier: FDA, IND)
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; GP160; BCG
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Single Usage / Single Dosage
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Assess for therapeutic biologics activity (proof-of-concept) (Experimental): Therapeutic Biological Product Mix activity - HIV GP160 0.1 mg x 1 mL add into BCG Organism 50 MG
  Interventions: Biological: HIV Therapeutic Biologic Mix - HIV GP160 plus BCG Vaccine Mix for percutaneous use

INTERVENTIONS:
Biological: HIV Therapeutic Biologic Mix - HIV GP160 plus BCG Vaccine Mix for percutaneous use — * By the percutaneous route with the multiple puncture device
  * HIV GP160 0.1 mg x 1 mL plus BCG Organism 50 MG Mix
  Other Names: GP160 plus BCG Vaccine Mix

SUMMARY:
Conducting an initial small, controlled clinical pharmacology trial to assess for therapeutic biologics activity (proof-of-concept) that suggests the potential for clinical benefit of HIV (+) patients

1. Treat Infection of Multiple Gene Mutation HIV Virus Strains.
2. Activate Human Antigen Presentation Reaction to HIV Specific Antigen.
3. The human antigen presenting cells (APCs) can take up and process HIV target antigen protein into small peptide fragments, and then HIV virus can be killed by APCs directly.

DETAILED DESCRIPTION:
* Conducting an initial small, controlled trial to assess therapeutic biologics activity (proof-of-concept) that suggests the potential for clinical benefit of HIV (+) patients without AIDS
* 20 HIV (+) patients with AIDS
* Positive HIV testing by standard RT-PCR assay or equivalent testing
* No symptoms of AIDS
* No clinical signs indicative of Severe or Critical Illness Severity
* HIV GP160 0.1 mg x 1 mL plus BCG Organism 50 MG Mix
* By the percutaneous route with the multiple puncture device
* Negative HIV testing by standard RT-PCR assay or equivalent testing after percutaneous use 3 weeks.
* Positive IGRA blood test with GP160 antigen after percutaneous use 21 days.
* Our trial duration will be up to 4 weeks.

ELIGIBILITY:
* Conducting an initial small, controlled trial to assess therapeutic biologics activity (proof-of-concept) that suggests the potential for clinical benefit of HIV (+) patients.
* 20 HIV (+) patients

Inclusion Criteria:

* HIV Positive
* Positive testing by standard RT-PCR assay or equivalent testing
* No AIDS Symptoms
* No clinical signs indicative of Severe or Critical Illness Severity
* Sign Informed Consent Form

Exclusion Criteria:

* Severe or Critical Illness Severity
* Pregnancy
* Breast-feeding
* The patients with other serious inter-current illness
* Serious Allergy
* Serious Bleed or Clot Tendency
* Serious side-effects of the biological product
* The prohibition of the biological product

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Number of HIV (+) Participants: | Duration up to 4 weeks
  * 20 HIV (+) patients
  * Positive HIV testing by standard RT-PCR assay
  * No AIDS Symptoms
  * No clinical signs indicative of Severe or Critical Illness Severity
Rate of Positive HIV nucleic acid: | Duration up to 4 weeks
  * 20 HIV (+) patients
  * Positive HIV testing by standard RT-PCR assay immediately
  * HIV nucleic acid testing, assessed by RT-PCR Assay Kit
  * Rate of Positive HIV nucleic acid must be 100%
Rate of Negative HIV nucleic acid: | Duration up to 4 weeks
  * 20 HIV (+) patients
  * HIV GP160 0.1 mg x 1 mL plus BCG Organism 50 MG Mix
  * By the percutaneous route with the multiple puncture device
  * Negative HIV by standard RT-PCR assay after percutaneous use 3 weeks
  * HIV nucleic acid testing, assessed by RT-PCR Assay Kit
  * Rate of Negative HIV nucleic acid will be more than 70%
20 HIV (+) Participants with IGRA blood test with HIV antigens | Duration up to 4 weeks
  - Positive IGRA blood test with HIV GP160 antigen after percutaneous use 3 weeks
20 HIV (+) Participants with IGRA blood test with TB antigens | Duration up to 4 weeks
  * Negative IGRA blood test with TB antigens before percutaneous use
  * Positive IGRA blood test with TB antigens after percutaneous use 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: HAN XU, MD/PhD/FAPCR, Study Chair — Medicine Invention Design Incorporation - IRB00009424; HAN XU, MD/PhD/FAPCR, Study Director — Medicine Invention Design Incorporation - IORG0007849; HAN XU, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design Incorporation - NPI 1023387701
Locations (1):
- Medicine Invention Design Incorporation - IORG0007849 - NPI 1023387701, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Netea MG, Dominguez-Andres J, Barreiro LB, Chavakis T, Divangahi M, Fuchs E, Joosten LAB, van der Meer JWM, Mhlanga MM, Mulder WJM, Riksen NP, Schlitzer A, Schultze JL, Stabell Benn C, Sun JC, Xavier RJ, Latz E. Defining trained immunity and its role in health and disease. Nat Rev Immunol. 2020 Jun;20(6):375-388. doi: 10.1038/s41577-020-0285-6. Epub 2020 Mar 4. PMID 32132681
- See also: FWA00015357 — http://ohrp.cit.nih.gov/search
- See also: IRB00009424 — http://ohrp.cit.nih.gov/search
- See also: IORG0007849 — http://ohrp.cit.nih.gov/search

DOCUMENTS (3):
  • Study Protocol (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT07182838/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT07182838/SAP_001.pdf
  • Informed Consent Form (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT07182838/ICF_002.pdf